CLINICAL TRIAL: NCT06415526
Title: Oncoplastic Entirely Robot-Assisted Approach (OPERA) - Incorporating Robotic Surgery in Both Mastectomy and DIEP Flap Reconstruction
Brief Title: OPERA - Incorporating Robotic Surgery in Both Mastectomy and DIEP Flap Reconstruction
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jung-Ju Huang, Associate Professor, Chang Gung Memorial Hospital
Other Study IDs: 202400581B0
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Mastectomy; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OPERA group: Patients with unilateral breast cancer received robotic-assisted mastectomy and robotic assisted free DIEP flap harvest for breast reconstruction
  Interventions: Procedure: OPERA

INTERVENTIONS:
Procedure: OPERA — Robotic-assisted mastectomy and robotic assisted free DIEP flap harvest for breast reconstruction

SUMMARY:
Current breast cancer surgery is achieving minimally invasive approach to reduce incision while providing better surgical vision and freedom in mastectomy. Breast reconstruction with free deep inferior epigastric artery perforator (DIEP) flap was considered the gold standard, however, the donor site morbidity remains an endless concern. Here we applied robotic-assisted surgery in both mastectomy and free DIEP flap harvest, so-called Oncoplastic Entirely Robot-Assisted Approach (OPERA).

A retrospective chart review identified 14 patients with unilateral breast cancer received robotic-assisted mastectomy and robotic assisted free DIEP flap harvest for breast reconstruction. The patient demographics and mastectomy and flap characteristics were reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA (American Society of Anesthesiologist) classification 1-2
* Breast skin should be free from cancer involvement, with adequate tumor to skin distance, and the largest preoperative tumor size no more than 5 cm
* The lesion should be located in any of the 4 quadrants away from the nipple, at least 1 cm distance between the lesion and the nipple

Exclusion Criteria:

* Patients with previous pelvis surgeries (except C-section)

Ages: 20 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with unilateral breast cancer received robotic-assisted mastectomy and robotic assisted free DIEP flap harvest for breast reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
ARS incision | Intra-operative
  The length of incision on anterior rectus sheath
Robotic time | Intra-operative
  The time it took to dissect pedicles with robotic arms
Flap size | Intra-operative
  The weight of the flap harvested

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuo WL, Wong AW, Tsai CY, Chen YF, Chang TN, Cheong DC, Huang JJ. Oncoplastic Entirely Robot-Assisted Approach: Incorporating Robotic Surgery in Both Mastectomy and DIEP Flap Reconstruction. Plast Reconstr Surg. 2025 Oct 1;156(4):451e-460e. doi: 10.1097/PRS.0000000000012157. Epub 2025 Apr 21. PMID 40261832